CLINICAL TRIAL: NCT05729386
Title: Phase 1 Study to Evaluate the Safety and the Pharmacokinetics of GC2129A in Healthy Adult Volunteers Under Fed Conditions
Brief Title: A Study to Evaluate the Safety, PK of GC2129A in Healthy Volunteers Under Fed Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: GC Biopharma Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GC2129A_BE_FED_P0102
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers
Keywords: PK; GC2129A
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Intervention Model Description: An open-label, randomized, fed, single-dose, 2-group, 2-period, crossover design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GC2129A + Reference drugs (Experimental): Period 1: GC2129A, Period 2: Individual Components
  Interventions: Drug: GC2129A(Period 1); Drug: Linaglptin 5mg and Metformin Hydrochloride 1000mg(Period 2)
- Reference drugs + GC2129A (Experimental): Period 1: Individual Components, Period 2: GC2129A
  Interventions: Drug: Linaglptin 5mg and Metformin Hydrocholoride 1000mg(Period 1); Drug: GC2129A(Period 2)

INTERVENTIONS:
Drug: GC2129A(Period 1) — Linagliptin and Metformin Hydrochloride Tablet
  Arms: GC2129A + Reference drugs
Drug: Linaglptin 5mg and Metformin Hydrocholoride 1000mg(Period 1) — Linagliptin 5mg/tab and Metformin Hydrochloride 1000mg/tab (2 tablets)
  Arms: Reference drugs + GC2129A
Drug: GC2129A(Period 2) — Linagliptin and Metformin Hydrochloride Tablet
  Arms: Reference drugs + GC2129A
Drug: Linaglptin 5mg and Metformin Hydrochloride 1000mg(Period 2) — Linagliptin 5mg/tab and Metformin Hydrochloride 1000mg/tab (2 tablets)
  Arms: GC2129A + Reference drugs

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics of oral administration of GC2129A in fed conditions to healthy adult volunteers.

DETAILED DESCRIPTION:
This study is an open-label, randomized, fasting, single-dose, 2-group, 2-period, crossover design to evaluate pharmacokinetics that are not affected by blinding. According to the order of administering the investigational drug for each period, 17 people are assigned to each of the two groups and administered.

For healthy subjects, each 17 subjects are assigned to each of the two groups(total 34 subjects). If the subject administrate GC2129A in the first period, the subject will be administrated reference drugs in the second period after washout(over 7 days). Conversely, if the subject administrate reference drugs in the first period, the subject will be administrated with GC2129A in the second period.

ELIGIBILITY:
Inclusion Criteria:

* A person who is 19 years of age or older at the time of a screening visit
* A person with a body mass index (BMI) of 18.0 kg/m2 or more and 30.0 kg/m2 or less with a weight of 50 kg or more (45 kg or more for women) during a screening visit
* A person who has no clinically significant congenital or chronic disease during a screening visit and has no pathological symptoms or findings as a result of internal examination

Exclusion Criteria:

* Persons with clinically significant diseases or history of the digestive system, cardiovascular system, endocrine system, respiratory system, blood and tumor, infectious disease, kidney and urinary reproductive system, mental and nervous system, musculoskeletal system, immune system, otolaryngology, skin system, and ophthalmology.
* A person who has a history of gastrointestinal surgery
* Those who have taken drug metabolism enzymes, such as barbiturate drugs, within one month of the first dose date or who have taken drugs that may interfere with this clinical trial within 10 days of the first dose date
* A person who participates in another clinical trial or biological equivalence test within six months of the first administration date
* A person who has donated whole blood within 8 weeks of the date of first administration, or has donated components within 2 weeks, or has received a blood transfusion within 4 weeks
* A person who is deemed unsuitable for participation in this clinical trial by the principle investigator(or the delegated sub-investigator) for reasons other than the above selection and exclusion criteria
* In the case of female volunteers, a pregnant woman or pregnant woman is suspected

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-04-17 (Estimated); Study Completion 2023-04-17 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) parameters - Cmax | 0-48hours
  Pharmacokinetic (PK) parameters of Metformin in serum
Pharmacokinetic (PK) parameters - AUCt | 0-48hours
  Pharmacokinetic (PK) parameters of Metformin in serum

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters - AUCinf | 0-48hours
  Pharmacokinetic (PK) parameters of Metformin in serum
Pharmacokinetic (PK) parameters - Tmax | 0-48hours
  Pharmacokinetic (PK) parameters of Metformin in serum
Pharmacokinetic (PK) parameters - t1/2 | 0-48hours
  Pharmacokinetic (PK) parameters of Metformin in serum

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus YangJi Hospital, Seoul, South Korea